CLINICAL TRIAL: NCT00003414
Title: Randomized Trial of Autologous GVHD for Refractory Lymphoma
Brief Title: Graft-Versus-Host Disease in Treating Patients With Recurrent or Refractory Lymphoma or Hodgkin's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: J9726 CDR0000066427; P30CA006973 (NIH); P01CA015396 (NIH); JHOC-97080106; JHOC-9726; NCI-V98-1453
Record Dates: First submitted 1999-11-01; First posted 2003-12-02 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-07

CONDITIONS: Graft Versus Host Disease; Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent/refractory childhood Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; graft versus host disease; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Graft vs Host Disease; Lymphoma; Hodgkin Disease; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — aldesleukin; Interferon-gamma; Busulfan; Cyclophosphamide; Cyclosporine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: aldesleukin
Biological: recombinant interferon gamma
Drug: busulfan
Drug: cyclophosphamide
Drug: cyclosporine
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Cyclosporine may induce graft-versus-host disease and make the body build an immune response that will kill cancer cells. Interleukin-2 and interferon gamma may enhance the effectiveness of graft-versus-host disease to kill cancer cells.

PURPOSE: Randomized phase III trial to determine the effectiveness of graft-versus-host disease in treating patients who have recurrent or refractory lymphoma or Hodgkin's disease .

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether autologous graft versus host disease significantly alters the relapse rate for lymphoma or Hodgkin's disease after autologous bone marrow transplantation.

OUTLINE: This is a randomized study. Stem cells are harvested and cryopreserved. All patients receive busulfan/cyclophosphamide or cyclosporine/total body irradiation as a preparative regimen. Arm I: Patients randomized to the graft versus host disease (GVHD) induction arm receive oral cyclosporine twice a day beginning on day 0 and continuing for at least 28 days, followed by peripheral blood stem cell (PBSC) infusion. At the time the white blood cell count begins to recover, subcutaneous interferon gamma is administered for 10 doses, followed 2 days later by subcutaneous interleukin-2 (IL-2) for 18 doses. Arm II: Patients do not receive autologous GVHD therapy after the PBSC transplant. Both arms should receive radiation to the site of lymphoma after recovering from the stem cell transplantation. Patients are followed at 6 months, 1 year, and 2 years posttransplant.

PROJECTED ACCRUAL: Approximately 50 patients (25 per arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Patients receiving autologous or syngeneic peripheral blood stem cell transplants for chemotherapy refractory or recurrent lymphoma or Hodgkin's disease, including: Progressive disease within 6 weeks of completing initial induction therapy OR Failure to achieve at least an overall partial response (at least a 50% reduction in tumor size) to conventional salvage therapy following relapse

PATIENT CHARACTERISTICS: Age: Any age Performance status: Not specified Life expectancy: Not specified Hematopoietic: No capillary leak syndrome Hepatic: Bilirubin no greater than 5 mg/dL Renal: Creatinine less than 4 mg/dL No renal failure requiring dialysis Cardiovascular: No hypotension No severe venooclusive disease Pulmonary: No pulmonary infiltrates OR No requirement for greater than 2 L oxygen Other: No weight gain greater than 5% of baseline weight No concurrent sepsis No temperature of 39 degrees C or higher for two or more days No clinically evident ascites

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Prior chemotherapy allowed Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 1997-10; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Relapse rate for lymphoma after autologous transplant | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Georgia B. Vogelsang, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Result] Bolanos-Meade J, Garrett-Mayer E, Luznik L, Anders V, Webb J, Fuchs EJ, Huff CA, Matsui W, Borrello IM, Brodsky R, Kasamon YL, Swinnen LJ, Flinn IW, Ambinder RF, Jones RJ, Hess AD, Vogelsang GB. Induction of autologous graft-versus-host disease: results of a randomized prospective clinical trial in patients with poor risk lymphoma. Biol Blood Marrow Transplant. 2007 Oct;13(10):1185-91. doi: 10.1016/j.bbmt.2007.06.011. Epub 2007 Aug 3. PMID 17889355